CLINICAL TRIAL: NCT00332202
Title: A Phase 3 Clinical Study to Investigate the Prevention of Relapse in Lymphoma Using Daily Enzastaurin
Brief Title: PRELUDE:Study to Investigate the Prevention of Relapse in Lymphoma Using Daily Enzastaurin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 9823; H6Q-MC-JCBJ (Other: Eli Lilly and Company); PRELUDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — enzastaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: enzastaurin
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily, until disease progression or maximum of 3 years
  Other Names: LY317615
  Arms: A
Drug: placebo — oral, daily
  Arms: B

SUMMARY:
This clinical research study is to investigate the prevention of relapse in patients with diffuse large B cell lymphoma (DLBCL) using enzastaurin daily.

This is a randomised trial which compares Enzastaurin to Placebo (dummy treatment), the chance of receiving Enzastaurin is 2 to 1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diffuse large B cell lymphoma
* Recently completed R-CHOP therapy and achieved remission
* International Prognostic Index (IPI) score 3,4,5
* At least 18 years of age
* Agree to study follow-up schedule

Exclusion Criteria:

* Have received therapy other than R-CHOP for lymphoma
* Serious medical condition such as infection,second cancer,heart disease
* Received radiation to more than one lesion
* Unable to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2006-06; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (153):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Robbinsdale, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Australia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gosford, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Casuarina, Northern Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prahran, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Belgium (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roeselare
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regina, Saskatchewan
- China (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suzhou
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herlev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki, Finland
- France (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Mans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chemnitz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari/Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aviano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Emilia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vicenza
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Col. Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toluca
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria da Feira
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hwasun-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hospitalet Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaragoza
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala
- Taiwan (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liouying/Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brighton, East Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maidstone, Kent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Crump M, Leppa S, Fayad L, Lee JJ, Di Rocco A, Ogura M, Hagberg H, Schnell F, Rifkin R, Mackensen A, Offner F, Pinter-Brown L, Smith S, Tobinai K, Yeh SP, Hsi ED, Nguyen T, Shi P, Hahka-Kemppinen M, Thornton D, Lin B, Kahl B, Schmitz N, Savage KJ, Habermann T. Randomized, Double-Blind, Phase III Trial of Enzastaurin Versus Placebo in Patients Achieving Remission After First-Line Therapy for High-Risk Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2016 Jul 20;34(21):2484-92. doi: 10.1200/JCO.2015.65.7171. Epub 2016 May 23. PMID 27217449
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzastaurin: Arm A - Experimental: Enzastaurin 500 milligram (mg) administered orally (PO) each day (QD) after an initial loading dose of 1125 mg on Day 1.
- Placebo: Arm B - Control: Placebo administered PO QD after an initial loading dose of placebo on Day 1.
Period: Overall Study
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Started | 504 | 254
Received At Least One Dose of Study Drug | 493 | 249
Completed | 263 | 129
Not Completed | 241 | 125
Not completed — Adverse Event | 72 | 28
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 6 | 8
Not completed — Protocol Entry Criteria Not Met | 6 | 5
Not completed — Protocol Violation | 7 | 2
Not completed — Sponsor Decision | 1 | 2
Not completed — Withdrawal by Subject | 36 | 17
Not completed — Progressive Disease | 106 | 60
Not completed — Death | 5 | 2

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT): All randomized participants.
Groups:
- Enzastaurin: Arm A - Experimental: Enzastaurin 500 mg administered PO QD after an initial loading dose of 1125 mg on Day 1.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control | Total
Number analyzed (Participants) | 504 | 254 | 758
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.19 (13.13) | 62.65 (12.09) | 62.35 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 105 | 350
  Male | 259 | 149 | 408
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 5 | 2 | 7
  Caucasian | 309 | 155 | 464
  East Asian | 144 | 73 | 217
  Hispanic | 24 | 13 | 37
  Native American | 1 | 0 | 1
  West Asian (Indian sub-continent) | 21 | 11 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 20 | 9 | 29
  Belgium | 10 | 4 | 14
  Brazil | 13 | 5 | 18
  Canada | 24 | 16 | 40
  China | 18 | 7 | 25
  Czechia | 6 | 2 | 8
  Germany | 15 | 10 | 25
  Denmark | 9 | 4 | 13
  Spain | 20 | 5 | 25
  Finland | 11 | 5 | 16
  France | 22 | 10 | 32
  Greece | 2 | 2 | 4
  Hungary | 4 | 2 | 6
  India | 22 | 11 | 33
  Italy | 15 | 10 | 25
  Japan | 54 | 33 | 87
  South Korea | 37 | 21 | 58
  Mexico | 13 | 9 | 22
  Poland | 9 | 7 | 16
  Puerto Rico | 3 | 1 | 4
  Portugal | 5 | 3 | 8
  Sweden | 19 | 5 | 24
  Taiwan | 24 | 8 | 32
  United Kingdom | 4 | 4 | 8
  United States | 125 | 61 | 186

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease-Free Survival
Description: Overall Disease-Free Survival (DFS) time is defined as the time from the date of study enrollment to the first date of objectively determined disease recurrence (progressive disease) or death from any cause. DFS was assessed according to International Working Group recommendations. Progressive disease (PD) is defined as a ≥ 50% increase from the lowest point in the sum of the product of the diameters (SPD) of any previously identified abnormal node for partial or nonresponders, or the appearance of any new lesion during or at the end of therapy.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (up to 80.30 months)
Population: All randomized participants. DFS is censored at the last assessable disease free assessment for participants who are alive or have not progressed. The number of censored participant data for enzastaurin and placebo is 369 (73.2%) and 180 (70.9%), respectively.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 504 | 254
Month | 42.8 [0.03 to 76.81] | 43.1 [0.03 to 80.30]
Statistical Analysis 1: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Test type: Superiority or Other; p = 0.541, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.689 to 1.216]

2. Secondary Outcome: Disease Free Survival at 2 Years
Description: Disease-free survival at 2 years (DFS2) is defined as the rate of DFS at 2 years from the date of study enrollment and is determined using the distribution of overall DFS times. Disease-free survival rates at 2 years will be estimated using the Kaplan-Meier method.
Time Frame: Baseline to 2 Years
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 504 | 254
proportion of participants | 0.785 [0.745 to 0.819] | 0.748 [0.687 to 0.798]

3. Secondary Outcome: Event-Free Survival
Description: Overall Event-Free Survival (EFS) time is defined as the time from the date of study enrollment to the first date of objectively determined disease recurrence (progressive disease), institution of a new anti-cancer treatment, or death from any cause. Progressive disease (PD) is defined as a ≥ 50% increase from the lowest point in the sum of the product of the diameters (SPD) of any previously identified abnormal node for partial or nonresponders, or the appearance of any new lesion during or at the end of therapy.
Time Frame: Baseline to Objective PD, Start of New Therapy or Death From Any Cause (up to 76.81 months)
Population: All randomized participants. EFS is censored at the last assessable disease-free assessment for participants who are alive, have not progressed or started new anticancer treatment. The number of censored participant data for enzastaurin and placebo is 364 (72.2%) and 176 (69.3%), respectively.
Measure: Number; unit: Month
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 504 | 254
Month
  Minimum EFS Survival | 0.03 | 0.03
  Maximum EFS Survival | 76.81 | 71.56

4. Secondary Outcome: Event-Free Survival at 2 Years
Description: Event-Free Survival at 2 years (EFS2) is defined as the rate of EFS at 2 years from the date of study enrollment and is determined using the distribution of overall EFS times. Event-free survival rates at 2 years will be estimated using the Kaplan-Meier method.
Time Frame: Baseline to 2 Years
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 504 | 254
Proportion of participants | 0.781 [0.741 to 0.816] | 0.734 [0.673 to 0.785]

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) time is defined as the time from the date of study enrollment to the date of death from any cause.
Time Frame: Baseline to Date of Death from Any Cause (up to 80.30 months)
Population: All randomized participants. Overall survival is censored at the last date of contact for participants who have no reported death. The number of censored participant data for enzastaurin and placebo is 404 (80.2%) and 205 (80.7%), respectively.
Measure: Number; unit: Month
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 504 | 254
Month
  Minimum OS Survival | 0.03 | 0.03
  Maximum OS Survival | 76.81 | 80.30

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of participants with treatment-emergent adverse events.
Time Frame: First dose through 30 days post-study treatment discontinuation (up to 81.30 months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 493 | 249
Participants | 459 | 230

7. Secondary Outcome: Quality of Life: Change From Baseline in Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Score
Description: The FACT-Lym assesses health-related quality of life (HRQoL) in participants with non-Hodgkin lymphoma. It includes the 27-item cancer-specific FACT-G (General), which assesses physical, social/family, emotional and functional well-being, plus a 15-item subscale that assesses concerns specific to lymphoma. Each item is scored on a scale from 0 (not at all) to 4 (very much), yielding a possible score of 0-168, with higher scores representing better HRQoL. This analysis utilized mixed-effect model repeated measure (MMRM) analysis of change from baseline adjusting for baseline covariates.
Time Frame: Baseline, Month 2; Baseline, Month 4; Baseline, Month 6; Baseline, Month 12; Baseline, Month 18; Baseline, Month 24; Baseline, Month 36
Population: All randomized participants who completed at least one FACT-Lym assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 348 | 189
Units on a Scale
  Month 2 | 2.45 (0.67) | 1.86 (0.93)
  Month 4 | 2.56 (0.80) | 2.51 (1.06)
  Month 6 | 2.04 (0.87) | 2.82 (1.10)
  Month 12 | 3.85 (0.87) | 2.11 (1.29)
  Month 18 | 2.87 (0.89) | 1.73 (1.26)
  Month 24 | 2.72 (0.99) | 3.96 (1.26)
  Month 36 | 2.54 (1.13) | 4.22 (1.43)
Statistical Analysis 1: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 2; Test type: Superiority or Other; p = 0.606, Mixed Models Analysis
Statistical Analysis 2: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 4; Test type: Superiority or Other; p = 0.971, Mixed Models Analysis
Statistical Analysis 3: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 6; Test type: Superiority or Other; p = 0.580, Mixed Models Analysis
Statistical Analysis 4: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 12; Test type: Superiority or Other; p = 0.265, Mixed Models Analysis
Statistical Analysis 5: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 18; Test type: Superiority or Other; p = 0.460, Mixed Models Analysis
Statistical Analysis 6: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 24; Test type: Superiority or Other; p = 0.441, Mixed Models Analysis
Statistical Analysis 7: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 36; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in EuroQol-5D (EQ-5D) Score
Description: The EQ-5D instrument is a participant-rated questionnaire used to evaluate health status. The EQ-5D assesses five dimensions (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression) that participants rate using three levels (no problem, some problem, or extreme problem), as well as overall health status. The five dimensions can be combined using country-specific weights to create an estimate of overall health status score. The possible values for score range from -0.594 (severe problems in all 5 dimensions) to 1 (no problem in all dimensions) on a scale where 1 represents the best possible health state. This analysis utilized mixed-effect model repeated measure (MMRM) analysis of change from baseline in the EQ-5D for the United Kingdom population-based index score adjusting for baseline covariates.
Time Frame: Baseline, Month 6; Baseline, Month 24; Baseline, Month 33
Population: All randomized participants who completed at least one EQ-5D assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Number analyzed (Participants) | 346 | 187
Units on a Scale
  Month 6 | 0.02 (0.01) | 0.00 (0.01)
  Month 24 | 0.02 (0.01) | 0.03 (0.02)
  Month 33 | 0.03 (0.01) | 0.03 (0.01)
Statistical Analysis 1: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 6; Test type: Superiority or Other; p = 0.267, Mixed Models Analysis
Statistical Analysis 2: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 24; Test type: Superiority or Other; p = 0.807, Mixed Models Analysis
Statistical Analysis 3: Comparison: Enzastaurin: Arm A - Experimental vs Placebo: Arm B - Control; Analysis for Month 33; Test type: Superiority or Other; p = 0.864, Mixed Models Analysis

9. Secondary Outcome: Translational Research: DFS Participants With Diffuse Large B-cell Lymphoma (DLBCL) Germinal-center B-cells (GCB) Versus Non-germinal-center B-cells
Description: Reported are the DFS for GCB and non-GCB status. DLBCL molecular subtypes of GCB/non-GCB using Hans' algorithm were determined by protein expression by immunohistochemistry (IHC) staining was used to assess molecular subtype characterization of GCB and non-GCB.
Time Frame: Baseline to 24 months (2 years)
Population: All randomized participants for which a pre-treatment tumor tissue was provided and had evaluable samples.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enzastaurin: Arm A - Experimental With Germinal-center B-cells: Enzastaurin 500 mg administered PO QD after an initial loading dose of 1125 mg on Day 1.Participants from enzastaurin treatment group with diffuse large B-cell lymphoma expression profile similar to germinal-center B-cells.
- Enzastaurin: Arm A - Experimental Non-germinal-center B-cells: Enzastaurin 500 mg administered PO QD after an initial loading dose of 1125 mg on Day 1. Participants from the placebo treatment group with diffuse large B-cell lymphoma expression profile not similar to germinal-center B-cells
- Placebo: Arm B - Control With Germinal-center B-cells: Placebo administered PO QD after an initial loading dose of placebo on Day 1.Participants from the placebo treatment group with diffuse large B-cell lymphoma expression profile not similar to germinal-center B-cells.
- Placebo Arm B- Control With Non-germinal-center B-cells: Placebo administered PO QD after an initial loading dose of placebo on Day 1. Participants from the placebo treatment group with diffuse large B-cell lymphoma expression profile not similar to germinal-center B-cells.
Arm/Group | Enzastaurin: Arm A - Experimental With Germinal-center B-cells | Enzastaurin: Arm A - Experimental Non-germinal-center B-cells | Placebo: Arm B - Control With Germinal-center B-cells | Placebo Arm B- Control With Non-germinal-center B-cells
Number analyzed (Participants) | 79 | 63 | 30 | 39
percentage of participants | 76.31 [65.1 to 84.4] | 75.97 [63.3 to 84.8] | 66.21 [46.3 to 80.2] | 68.20 [50.7 to 80.6]
Statistical Analysis 1: Comparison: Enzastaurin: Arm A - Experimental With Germinal-center B-cells vs Enzastaurin: Arm A - Experimental Non-germinal-center B-cells; Test type: Superiority; p = 0.400, Regression, Cox; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.415 to 1.420]
Statistical Analysis 2: Comparison: Placebo: Arm B - Control With Germinal-center B-cells vs Placebo Arm B- Control With Non-germinal-center B-cells; Test type: Superiority; p = 0.539, Regression, Cox; Hazard Ratio (HR) = 1.309, 95% CI 2-sided [0.557 to 3.080]

10. Secondary Outcome: Translational Research: DFS of Participants With Diffuse Large B-cell Lymphoma (DLBCL) Protein Kinase C-β2 (PKC-β2) Expression
Description: Reported are the DFS based on PKC-β2 protein expression. Immunohistochemistry (IHC) staining was performed to assess protein expression of PKC-β2 in cytoplasm scored for percent of tumor cells stained, and using 50% positive staining as the cutoff for high/low expression (high expression: >=50% staining, low expression: <50% staining).
Time Frame: Baseline to 94.5 months
Population: All randomized participants for which a pre-treatment tumor tissue was provided and had evaluable samples.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enzastaurin: Arm A With PKC-β2 Cytoplasm (High Expression); Enzastaurin: Arm A With PKC-β2 Cytoplasm (Low Expression): Participants from enzastaurin treatment groups with PKC-β2 cytoplasmic protein expression.
- Placebo: Arm B With PKC-β2 Cytoplasm (High Expression); Placebo: Arm B With PKC-β2 Cytoplasm (Low Expression): Participants from placebo treatment group with PKC-β2 cytoplasmic protein expression.
Arm/Group | Enzastaurin: Arm A With PKC-β2 Cytoplasm (High Expression) | Enzastaurin: Arm A With PKC-β2 Cytoplasm (Low Expression) | Placebo: Arm B With PKC-β2 Cytoplasm (High Expression) | Placebo: Arm B With PKC-β2 Cytoplasm (Low Expression)
Number analyzed (Participants) | 39 | 117 | 21 | 50
percentage of participants | 64.86 [47.3 to 77.9] | 81.16 [72.6 to 87.3] | 61.54 [37.6 to 78.6] | 70.58 [55.3 to 81.5]
Statistical Analysis 1: Comparison: Enzastaurin: Arm A With PKC-β2 Cytoplasm (High Expression) vs Placebo: Arm B With PKC-β2 Cytoplasm (High Expression); Test type: Superiority or Other; p = 0.084, Regression, Cox; Hazard Ratio (HR) = 1.775, 95% CI 2-sided [0.947 to 3.329]
Statistical Analysis 2: Comparison: Enzastaurin: Arm A With PKC-β2 Cytoplasm (Low Expression) vs Placebo: Arm B With PKC-β2 Cytoplasm (Low Expression); Test type: Superiority; p = 0.585, Regression, Cox; Hazard Ratio (HR) = 1.286, 95% CI 2-sided [0.527 to 3.137]

11. Secondary Outcome: Pharmacokinetics: Average Steady-State Concentration (Cavg,ss) for Total Analyte
Time Frame: Month 2, Month 4: Predose
Population: All participants who received at least one dose of the study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Groups:
- Total Enzastaurin Population: All participants who received enzastaurin 500 mg PO QD after an initial loading dose of 1125 mg on Day 1.
Arm/Group | Total Enzastaurin Population
Number analyzed (Participants) | 328
nanomole/liter (nmol/L) | 2370 (59.9)

ADVERSE EVENTS:
Groups:
- Enzastaurin: Arm A - Experimental: Administered orally as four 125-mg tablets daily (after an initial loading dose of three 125-mg tablets given three times on Day 1)
- Placebo: Arm B - Control: Administered orally as four tablets daily (after an initial loading dose of three tablets given three times on Day 1)
Arm/Group | Enzastaurin: Arm A - Experimental | Placebo: Arm B - Control
Serious Adverse Events (participants affected / at risk) | 135/493 | 72/249
Other Adverse Events (participants affected / at risk) | 406/493 | 185/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin: Arm A - Experimental (N=493) | Placebo: Arm B - Control (N=249)
Anaemia (Blood and lymphatic system disorders) | 5 (9) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (15)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (11) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (3)
Cardiac failure (Cardiac disorders) | 3 (16) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 2 (4)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 3 (25) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (6) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (3)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (8) | 0 (0)
Cataract (Eye disorders) | 2 (4) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (2) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (5) | 1 (6)
Ophthalmoplegia (Eye disorders) | 0 (0) | 1 (2)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (17)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (13) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis ulcerative (Gastrointestinal disorders) | 1 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 1 (11) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 1 (1)
Pseudopolyposis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (15)
Asthenia (General disorders) | 2 (4) | 1 (2)
Chest pain (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (2) | 0 (0)
Multi-organ disorder (General disorders) | 0 (0) | 1 (3)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 0 (0)
Spinal pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (6) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (7) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (2) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Cervicitis (Infections and infestations) | 1/239 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 2 (3)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 1 (2)
Hepatitis b (Infections and infestations) | 0 (0) | 3 (11)
Hepatitis c (Infections and infestations) | 1 (7) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (11) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Myelitis (Infections and infestations) | 0 (0) | 1 (10)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 7 (10)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Scrub typhus (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (7) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5) | 0 (0)
Urosepsis (Infections and infestations) | 2 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (12) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 2/239 (8) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (7) | 1 (17)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (10)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (3)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 3 (12) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (21)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (9) | 1 (14)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (9) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (10)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (7) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (6) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/239 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/254 (5) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (9) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (18) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve paralysis (Nervous system disorders) | 0 (0) | 1 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (6)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2)
Grand mal convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (15)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (15)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 (4) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (9)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (3) | 1 (3)
Syncope (Nervous system disorders) | 6 (8) | 0 (0)
Tongue paralysis (Nervous system disorders) | 0 (0) | 1 (15)
Tonic convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (3)
Vith nerve paralysis (Nervous system disorders) | 1 (2) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (14) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (6) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (3) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (4) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1/254 (12) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1/254 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (23) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (8) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 1 (2) | 0 (0)
Anal fissure excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (9) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (21) | 0 (0)
Hypotension (Vascular disorders) | 1 (4) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin: Arm A - Experimental (N=493) | Placebo: Arm B - Control (N=249)
Anaemia (Blood and lymphatic system disorders) | 33 (221) | 13 (79)
Leukopenia (Blood and lymphatic system disorders) | 27 (87) | 11 (45)
Neutropenia (Blood and lymphatic system disorders) | 52 (143) | 26 (66)
Abdominal pain (Gastrointestinal disorders) | 40 (140) | 12 (20)
Constipation (Gastrointestinal disorders) | 49 (256) | 20 (101)
Diarrhoea (Gastrointestinal disorders) | 97 (387) | 33 (115)
Dry mouth (Gastrointestinal disorders) | 25 (177) | 5 (44)
Faeces discoloured (Gastrointestinal disorders) | 39 (340) | 0 (0)
Nausea (Gastrointestinal disorders) | 73 (195) | 38 (150)
Vomiting (Gastrointestinal disorders) | 47 (64) | 26 (44)
Fatigue (General disorders) | 91 (628) | 45 (304)
Oedema peripheral (General disorders) | 63 (370) | 16 (84)
Pyrexia (General disorders) | 34 (60) | 16 (21)
Nasopharyngitis (Infections and infestations) | 37 (112) | 13 (34)
Upper respiratory tract infection (Infections and infestations) | 42 (80) | 15 (47)
Urinary tract infection (Infections and infestations) | 27 (93) | 7 (13)
Alanine aminotransferase increased (Investigations) | 27 (148) | 12 (73)
Aspartate aminotransferase increased (Investigations) | 29 (191) | 12 (52)
Electrocardiogram qt prolonged (Investigations) | 54 (317) | 11 (44)
Weight increased (Investigations) | 24 (194) | 19 (149)
Decreased appetite (Metabolism and nutrition disorders) | 34 (151) | 14 (56)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (368) | 28 (238)
Back pain (Musculoskeletal and connective tissue disorders) | 52 (353) | 24 (213)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 (263) | 15 (107)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 (173) | 17 (71)
Dizziness (Nervous system disorders) | 53 (238) | 21 (129)
Headache (Nervous system disorders) | 49 (295) | 32 (189)
Insomnia (Psychiatric disorders) | 40 (327) | 13 (107)
Chromaturia (Renal and urinary disorders) | 96 (916) | 1 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 76 (283) | 30 (130)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 (84) | 7 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 51 (329) | 21 (104)
Rash (Skin and subcutaneous tissue disorders) | 56 (323) | 27 (120)
Hypertension (Vascular disorders) | 8 (64) | 13 (127)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days